CLINICAL TRIAL: NCT02171858
Title: Multivariate Analysis of Serum High Sensitivity C-Reactive Protein in Patients With Acute Phase Stroke
Acronym: MAASP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Central Sur de Alta Especialidad (Other)
Responsible Party: Principal Investigator, Jorge Yanez, Md, Hospital Central Sur de Alta Especialidad
Other Study IDs: CRP-S1
Record Dates: First submitted 2014-06-04; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Stroke; National Institutes of Health Stroke Scale; Serum High Sensitivity C-Reactive Protein
Keywords: Stroke; National Institutes of Health Stroke Scale; Serum high sensitivity C-Reactive Protein
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- stroke: Patients admitted to hospital who are diagnosed with stroke will be treated as usually a our center by observation, venous or arterial thrombolysis depending on extension, condition, thrombolysis feasibility.

SUMMARY:
Stroke is one of main causes of death and impairment worldwide. Objective of this study is to analyze serum High Sensitivity C-Reactive Protein in acute phase stroke in patients attended at Petróleos Mexicanos Hospital Central Sur de Alta Especialidad and to correlate with stroke extension and clinical features.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of acute phase stroke who arrive to emergency room at our hospital
* Patients affiliated to Petróleos Mexicanos medical system
* Patients of any gender
* Patients between 18 and 80 years old

Exclusion Criteria:

* Stroke provoked by angiographic procedure
* Pregnancy
* Patient under chemotherapy or radiotherapy
* Recently surgery or trauma among last 30 days
* Heparin usage
* Stroke and/ or thrombolysis history
* Active infection
* Liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affiliated to Petróleos Mexicanos medical system of any gender between 18 and 80 years old suspected of acute phase stroke who arrive to emergency room at our hospital
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Measure of serum High sensitivity C-Reactive Protein level | within the first 8 hours since admission to hospital
  Serum levels of serum High sensitivity C-Reactive Protein will be measured in patients with suspicion of stroke at the emergency room within the first 8 hours of arrival at our hospital

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale | within the first 4 hours since admission to emergency room
  clinical impact of stroke will be determined by neurology and neurosurgery department at admission to emergency room of our hospital

OTHER OUTCOMES:
Stroke extension | within the first 4 hours since admission to emergency room
  brain image will be taken as soon as possible when patient suspected with stroke arrives to emergency room and after clinical evaluation
Origin of stroke | origin will be diagnosed during the hospital stay expecting no more than 1 week
  origin of stroke will be investigated within hospital stay
Hospital stay | hospital stay is expected for no more than 1 week unless intensive care unit is needed
  from arrival of patient to emergency room until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Central Sur Alta Especialidad, Mexico City, Tlalpan, Mexico